CLINICAL TRIAL: NCT02177487
Title: An Open-Label, Six Month Safety Evaluation of the Fixed Dose Combination of Telmisartan 80 mg Plus Hydrochlorothiazide 12.5 mg in Patients With Mild-to-Moderate Hypertension
Brief Title: Safety Evaluation of Telmisartan Plus Hydrochlorothiazide in Patients With Mild-to-Moderate Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 502.321
Record Dates: First submitted 2014-06-26; First posted 2014-06-27 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — telmisartan, hydrochlorothiazide drug combination

ARMS (1):
- Telmisartan + Hydrochlorothiazide (Experimental)
  Interventions: Drug: Telmisartan/hydrochlorothiazide

INTERVENTIONS:
Drug: Telmisartan/hydrochlorothiazide

SUMMARY:
Study to assess the safety of six month of open-label, treatment with the fixed dose combination of telmisartan 80 mg plus hydrochlorothiazide 12.5 mg in a subset of patients with mild-to-moderate hypertension who completed the eight week randomized, double blind 502.261 study.

ELIGIBILITY:
Inclusion Criteria:

* All patients who were randomized and completed all study visits of the preceding double-blind trial with the fixed dose combination (502.261) who meet the following criteria:

  * Patients that are not controlled on telmisartan 80 mg monotherapy at the final visit (Visit 6) of the 502.261 study
* Patients who are able to provide written informed consent
* Patients who are able to enter the study immediately upon their completion of the preceding double-blind trial of the fixed dose combination (502.261)

Exclusion Criteria:

* Patients with any exclusion criterion (except criteria 1, 19 and 20), as defined in the preceding study (502.261):

  * Pre-menopausal women (last menstruation ≤ 1 year prior to start of screening)

    * who are not surgically sterile (hysterectomy, tubal ligation)
    * who are NOT practicing acceptable means of birth control or who do NOT plan to continue using an acceptable method throughout the study. Acceptable methods of birth control include intrauterine device (IUD), oral, implantable or injectable contraceptives
  * Any women:

    * who has a positive serum pregnancy test at screening (Visit 1) or baseline (Visit 4)
    * who has a positive urine pregnancy test prior to taking the first dose of open-label medication (at Visit 2)
    * who is nursing
  * Hepatic and/or renal dysfunction as defined by the following laboratory parameters:

    * SGPT (ALT) (serum glutamate pyruvate transaminase) or SGOT (AST) (serum glutamate oxaloacetate transaminase) greater than two times the upper limit of normal
    * Serum creatinine > 2.3 mg/dL
  * Clinically relevant sodium depletion, hyperkalemia, or hypokalemia at baseline
  * Known or suspected secondary hypertension
  * Bilateral renal artery stenosis; renal artery stenosis in a solitary kidney; post-renal transplant patients, presence of only one functioning kidney
  * Congestive heart failure (CHF) (NYHA (New York Heart Association) class CHF III-IV)
  * Unstable angina within the past three months
  * Stroke within the past six months
  * Myocardial infarction or cardiac surgery within the past three months
  * PTCA (percutaneous transluminal coronary angioplasty) within the past three months
  * History of angioedema
  * Sustained ventricular tachycardia, atrial fibrillation, atrial flutter or other clinically relevant cardiac arrhythmias as determined by the investigator
  * Hypertrophic obstructive cardiomyopathy, aortic stenosis, hemodynamically relevant stenosis of the aortic or mitral valve
  * Administration of digoxin or other digitalis-type drugs
  * Patients with insulin treated Type II diabetes mellitus whose diabetes has not been stable and controlled for at least the past three months as defined by an HbA1C ≥ 10%
  * Known drug or alcohol dependency within the past one year period
  * Known hypersensitivity to any component of the formulations
  * Any clinical condition which, in the opinion of the investigator, would not allow safe completion of the protocol and safe administration of trial medication

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 1999-06; Primary Completion 2000-01 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | up to 6 months
Changes from baseline in laboratory tests | Baseline and month 6
Changes from baseline in physical examination | Baseline and month 6
Changes from baseline in 12-lead ECG (electrocardiogram) | Baseline and month 6
Changes from baseline in seated blood pressure | Baseline, month 1, 3 and 6
Changes from baseline in pulse rate | Baseline, month 1, 3 and 6